CLINICAL TRIAL: NCT02099331
Title: Cardiac Surgery and the Risk of Atrial Fibrillation: an Intervention Trial Evaluating Melatonin
Acronym: DREAM
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of faculty staffing
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NA_00090647
Record Dates: First submitted 2014-03-22; First posted 2014-03-28 (Estimated); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Reactive Oxygen Species; Cardiac Surgery
MeSH Terms: conditions — Atrial Fibrillation | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Experimental): The investigators will administer melatonin at 40mg by mouth (two 20 mg tablets), nightly prior to sleep. The administration will start 2 days prior to the scheduled surgery date and will continue until post-operative day 3.
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): The investigators will administer matching Placebo by mouth (two tablets to match Melatonin), nightly prior to sleep. The administration will start 2 days prior to the scheduled surgery date and will continue until post-operative day 3.
  Interventions: Drug: Placebo (for Melatonin)

INTERVENTIONS:
Drug: Melatonin
  Other Names: N - acetyl - 5 - methoxytryptamine
  Arms: Melatonin
Drug: Placebo (for Melatonin) — Sugar pill manufactured to mimic Melatonin 20 mg
  Arms: Placebo

SUMMARY:
Atrial fibrillation is a common heart rhythm condition that can occur after cardiac surgery and has been associated with an increase in hospital length of stay, overall hospital costs, worsening clinical condition and higher rates of death. Newer research indicates that inflammation is a key contributor to atrial fibrillation in this setting.

Melatonin is a naturally made hormone that is regarded as an extremely effective anti-inflammatory substance, with a very favorable safety profile. This clinical trial is being done to test the ability of melatonin to reduce the risk of developing atrial fibrillation after cardiac surgery.

This is a research study where patients will be given either oral melatonin at 40 mg or placebo nightly prior to sleep. The study product will start approximately 2 days prior to the scheduled surgery date and will continue until the 3rd day after the operation. The remainder of the clinical care will remain the same.

The investigators project that patients who receive melatonin will have a significant decrease in the occurrence of atrial fibrillation after surgery.

DETAILED DESCRIPTION:
Atrial fibrillation is the most common arrhythmia to occur after coronary artery bypass graft (CABG) surgery. This arrhythmia occurs in approximately 1 in every 3 patients in this setting and the rate is even higher after valve or combined valve and CABG procedures. The majority of episodes of atrial fibrillation occur within the first 3 days after cardiac surgery and for those who have an initial episode of atrial fibrillation, the majority will go on to have another recurrence within 2 days of the first episode. Postoperative atrial fibrillation has been associated with an increase in neurological, renal and infectious complications as well as prolonged hospitalization and a significant increase in overall healthcare costs.

There is a considerable amount of emerging data indicating that inflammation and oxidative stress, by way of reactive oxygen species (ROS), associated with cardiac surgery and cardiopulmonary bypass (CPB) may play an important role in the in the development of postoperative atrial fibrillation. Prior animal studies have demonstrated that ROS may lead to electroanatomical remodeling and increase the vulnerability to atrial fibrillation by promoting progressive fibrosis and subsequent alteration of the extracellular matrix. A few randomized controlled trials have demonstrated the beneficial effects of pre-treatment with anti-inflammatory medications such as statins for the prevention of post-operative atrial fibrillation. With this in mind, other anti-inflammatory therapies may also be effective in preventing postoperative atrial fibrillation.

Melatonin (N - acetyl - 5 - methoxytryptamine) is the main product secreted from the pineal gland and has been shown to be a powerful scavenger of ROS and is regarded as the most potent endogenous antioxidant. In fact, melatonin is more effective than other antioxidants in removing free radicals and it has both lipophilic and hydrophilic properties contributing to its more consistent penetration through cellular membranes. In addition to being a naturally synthesized hormone, melatonin has been shown to have a very favorable safety profile when administered in the clinical setting.

For these reasons, investigators have designed a randomized, double-blind, placebo-controlled trial where patients who are to undergo cardiac surgery and CPB, will be randomized to melatonin or placebo and the investigators will determine the incidence of post operative atrial fibrillation in both groups. Additionally, the investigators will measure ROS from serum as well as right atrial appendage samples of subjects and assess the effects of melatonin on ROS levels as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Age over the age of 18.
2. Scheduled for elective cardiac surgery (coronary artery bypass grafting, valvular surgery or combined procedures)
3. Enroll at least 48 hours before surgery is scheduled
4. Presence of normal sinus rhythm on screening electrocardiogram.
5. Be willing to provide informed consent (which may be provided by a legally authorized representative if the patient is not able to do so).

Exclusion Criteria:

1. History of prior atrial fibrillation
2. Inability to give informed consent.
3. Use of anti-arrhythmic drugs other than beta-blockers
4. Chronic NSAID or antioxidant use
5. History of severe autoimmune disorders with the need for autoimmune medications.
6. History of epilepsy.
7. Compromised hepatic function (aminotransferase levels > 1.5 times the upper limit of normal)
8. Current pregnancy (determined by either serum or urine pregnancy test, as ordered by the primary team)
9. Non-English Speakers
10. Current use of warfarin, nifedipine, fluvoxamine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-07-06 (Actual); Study Completion 2015-07-06 (Actual)

PRIMARY OUTCOMES:
Incidence of atrial fibrillation | 2 years
  At the end of the study, the primary outcome of incident atrial fibrillation will be assessed in each study arm.

SECONDARY OUTCOMES:
Levels of Reactive Oxygen Species (ROS) | 2 years
  The investigators will measure levels of ROS from the right atrial appendage and serum samples at the time of surgery as well as on a daily basis from the serum for three days after surgery. Specifically, the investigators will measure NADPH oxidase, peroxide anion, peroxynitrite and thiobarbituric acid reactive substances. At the end of the study, the investigators will compare these levels in both arms.

OTHER OUTCOMES:
Adverse Events | 2 years
  The investigators will measure the incidence of MACE (need for redo surgery, acute heart failure, death or malignant arrhythmias) as well hepatic dysfunction and renal failure in each arm of the study.
Impact on Sleep | 2 years
  The investigators will measure how the intervention may impact the amount of sleep patients attain in the first 72 hours after surgery. This outcome measure will be compared between the arms at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Cingolani, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States